CLINICAL TRIAL: NCT04602598
Title: A Phase II, Single-Site, Open-Label Study of Zanubrutinib in Patients With IgG4-Related Disease
Brief Title: Zanubrutinib in Patients With IgG4-Related Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Matthew C. Baker (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor-Investigator, Matthew C. Baker, Assistant Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 58497
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: IgG4 Related Disease
MeSH Terms: conditions — Immunoglobulin G4-Related Disease | interventions — zanubrutinib

STUDY DESIGN:
Intervention Model Description: Open-label study in symptomatic subjects with histopathologically confirmed IgG4-related disease affecting the submandibular and/or lacrimal glands. Ten subjects will be included in the study. All eligible subjects will receive zanubrutinib 80mg BID over a period of 24 weeks and will be followed up for an additional 8 weeks after the last dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Zanubrutinib (Experimental): Zanubrutinib orally at a dose of 80mg BID for 24 weeks
  Interventions: Drug: Zanubrutinib 80 MG

INTERVENTIONS:
Drug: Zanubrutinib 80 MG — Zanubrutinib 80 MG for 24 weeks

SUMMARY:
The aim of this clinical trial is to evaluate the safety and efficacy of zanubrutinib in treating patients with IgG4-related disease

DETAILED DESCRIPTION:
This will be a single-site, open-label study in symptomatic patients with IgG4-related disease affecting the submandibular and/or lacrimal glands. All patients will receive zanubrutinib orally at a dose of 80mg BID for 24 weeks.

The primary objective of this study is to demonstrate that zanubrutinib treatment reduces reduces the volume of the submandibular and/or lacrimal glands on PET/MRI at week 24 compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 to 85, inclusive, at the time of initial screening
* Have histopathologically confirmed IgG4-RD in the submandibular gland and/or the lacrimal gland confirmed by international consensus pathology criteria

  * Presence of a lymphoplasmacytic infiltrate with 10 IgG4+ plasma cells per high-power field and/or an IgG4+/IgG+ plasma cell ratio of 40%
* All women must test negative for pregnancy and agree to use a reliable method of birth control
* No current treatment with immunosuppressive medications other than prednisone 40mg daily (or other glucocorticoid equivalent) with stable dosing for 28 days

Exclusion Criteria:

* Unstable prescribed dose of glucocorticoids within 28 days prior to baseline
* Any treatment with a synthetic DMARD including but not limited to hydroxychloroquine, methotrexate, leflunomide, or sulfasalazine within 28 days prior to baseline
* Any treatment with a cytotoxic or immunosuppressive drug including but not limited to cyclophosphamide, mycophenolic acid, azathioprine, cyclosporine, sirolimus, or tacrolimus within 28 days prior to baseline
* Any treatment with a BTK inhibitor within 6 months before baseline
* Any treatment with a JAK inhibitor within 28 days prior to baseline
* Use of biologic agents including infliximab, abatacept, or tocilizumab within 56 days prior to baseline
* Use of a B cell depleting therapy (such as rituximab) within 12 months prior to baseline
* A history of, or current, inflammatory or autoimmune disease (that could affect the interpretation of safety or efficacy outcomes) other than IgG4-related disease
* Evidence of active tuberculosis, HIV, or hepatitis B or C infection
* History of cancer other than non-melanoma skin cancer, cervical dysplasia or carcinoma in situ (cured >1 year), prostate cancer (cured >5 years), or colon cancer (cured >5 years)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Volume of the submandibular glands on PET-MRI | Baseline to Week 24
  To demonstrate that zanubrutinib treatment reduces the volume of the submandibular glands on PET-MRI at Week 24 compared to Baseline.
Volume of the lacrimal glands on PET-MRI | Baseline to Week 24
  To demonstrate that zanubrutinib treatment reduces the volume of the lacrimal glands on PET-MRI at Week 24 compared to Baseline.

SECONDARY OUTCOMES:
FDG avidity (SUVmax) of the submandibular glands on PET | Baseline to Week 24
  Effect of zanubrutinib on change in FDG avidity (SUVmax) of the submandibular glands on PET at Week 24 compared to Baseline.
FDG avidity (SUVmax) of the lacrimal glands on PET | Baseline to Week 24
  Effect of zanubrutinib on change in FDG avidity (SUVmax) of the lacrimal glands on PET at Week 24 compared to Baseline.
Change in metabolic lesion volume (MLV) of submandibular and/or lacrimal glands on PET | Baseline to Week 24
Change in total lesion glycolysis (TLG) of submandibular and/or lacrimal glands on PET | Baseline to Week 24
Change in submandibular glands on MRI | Baseline to Week 24
  Change in parenchymal architecture scored 0 to 4 and sialography scored 0 to 4
Change in parotid glands on MRI | Baseline to Week 24
  Change in parenchymal architecture scored 0 to 4 and sialography scored 0 to 4
Change in lacrimal glands on MRI | Baseline to Week 24
  Change in parenchmyal architecture scored 0 to 4 and sialography scored 0 to 4
Change in the volume of the parotid glands on PET/MRI | Baseline to Week 24
Change in the volume of the submandibular glands on PET/MRI | Baseline to Week 12
Change in the volume of the lacrimal glands on PET/MRI | Baseline to Week 12
Change in the volume of the parotid glands on PET/MRI | Baseline to Week 12
FDG avidity (SUVmax) of the submandibular and/or lacrimal glands on PET | Baseline to Week 12
  Effect of zanubrutinib on change in FDG avidity (SUVmax) of the submandibular and/or lacrimal glands on PET at Week 12 compared to Baseline.
Change in metabolic lesion volume (MLV) of submandibular and/or lacrimal glands on PET | Baseline to Week 12
Change in total lesion glycolysis (TLG) of submandibular and/or lacrimal glands on PET | Baseline to Week 12
Change in submandibular glands on MRI | Baseline to Week 12
  Change in parenchymal architecture scored 0 to 4 and sialography scored 0 to 4
Change in parotid glands on MRI | Baseline to Week 12
  Change in parenchymal architecture scored 0 to 4 and sialography scored 0 to 4
Change in lacrimal glands on MRI | Baseline to Week 12
  Change in parenchmyal architecture scored 0 to 4 and sialography scored 0 to 4
Change in serum IgG4 level | Baseline to Week 24
Change in serum IgG4 level | Baseline to Week 12
Change in plasmablast count | Baseline to Week 24
Change in plasmablast count | Baseline to Week 12
Change in absolute regulatory B cell count | Baseline to Week 24
Change in absolute regulatory B cell count | Baseline to Week 12
Change in the IgG4-RD Responder Index | Baseline to Week 24
Change in the IgG4-RD Responder Index | Baseline to Week 12
Proportion of patients with no disease flares | Week 12 to Week 24
Change in total salivary grey scale ultrasound score (TUS) | Baseline to Week 24
  Each parotid and submandibular gland scored from 0 to 3 with a higher score indicating worse disease, total summed scores across all four glands will be assessed for change
Change in total salivary grey scale ultrasound score (TUS) | Baseline to Week 12
  Each parotid and submandibular gland scored from 0 to 3 with a higher score indicating worse disease, total summed scores across all four glands will be assessed for change
Change in highest score among the salivary glands for the grey scale ultrasound score (HSUS) | Baseline to Week 24
  Each parotid and submandibular gland scored from 0 to 3 with a higher score indicating worse disease, highest score will be assessed for change
Change in highest score among the salivary glands for the grey scale ultrasound score (HSUS) | Baseline to Week 12
  Each parotid and submandibular gland scored from 0 to 3 with a higher score indicating worse disease, highest score will be assessed for change
Change in glandular inflammation total ultrasound score (iTUS) | Baseline to Week 24
  Each parotid and submandibular gland scored from 0 to 3 with a higher score indicating worse disease, total summed scores across all four glands will be assessed for change
Change in glandular inflammation total ultrasound score (iTUS) | Baseline to Week 12
  Each parotid and submandibular gland scored from 0 to 3 with a higher score indicating worse disease, total summed scores across all four glands will be assessed for change
Change in highest score among the salivary glands for the glandular inflammation ultrasound score (iHSUS) | Baseline to Week 24
  Each parotid and submandibular gland scored from 0 to 3 with a higher score indicating worse disease, highest score will be assessed for change
Change in highest score among the salivary glands for the glandular inflammation ultrasound score (iHSUS) | Baseline to Week 12
  Each parotid and submandibular gland scored from 0 to 3 with a higher score indicating worse disease, highest score will be assessed for change
Change in physician global assessment of disease | Baseline to Week 24
  Symptoms rated on a 100 mm VAS. Score range: 0 to 100, higher scores correspond to worse disease state.
Change in physician global assessment of disease | Baseline to Week 12
  Symptoms rated on a 100 mm VAS. Score range: 0 to 100, higher scores correspond to worse disease state.
Change in patient global assessment of disease | Baseline to Week 24
  Symptoms rated on a 100 mm VAS. Score range: 0 to 100, higher scores correspond to worse disease state.
Change in patient global assessment of disease | Baseline to Week 12
  Symptoms rated on a 100 mm VAS. Score range: 0 to 100, higher scores correspond to worse disease state.
Change in VAS for ocular symptoms | Baseline to Week 24
  Symptoms rated on a 100 mm VAS. Score range: 0 to 100, higher scores correspond to worse disease state.
Change in VAS for ocular symptoms | Baseline to Week 12
  Symptoms rated on a 100 mm VAS. Score range: 0 to 100, higher scores correspond to worse disease state.
Change in VAS for salivary symptoms | Baseline to Week 24
  Symptoms rated on a 100 mm VAS. Score range: 0 to 100, higher scores correspond to worse disease state.
Change in VAS for salivary symptoms | Baseline to Week 12
  Symptoms rated on a 100 mm VAS. Score range: 0 to 100, higher scores correspond to worse disease state.
Change in FACIT-F fatigue score | Baseline to Week 24
  Total score range: 0-52, lower scores correspond with more fatigue.
Change in FACIT-F fatigue score | Baseline to Week 12
  Total score range: 0-52, lower scores correspond with more fatigue.
Change in RAND Short Form-36 | Baseline to Week 24
Change in RAND Short Form-36 | Baseline to Week 12
Change in C3 lab | Baseline to Week 24
Change in C3 lab | Baseline to Week 12
Change in C4 lab | Baseline to Week 24
Change in C4 lab | Baseline to Week 12
Change in total IgG lab | Baseline to Week 24
Change in total IgG lab | Baseline to Week 12
Change in IgE lab | Baseline to Week 24
Change in IgE lab | Baseline to Week 12
Change in IgG1 lab | Baseline to Week 24
Change in IgG1 lab | Baseline to Week 12
Change in ESR lab | Baseline to Week 24
Change in ESR lab | Baseline to Week 12
Change in CRP lab | Baseline to Week 24
Change in CRP lab | Baseline to Week 12
Incidence of safety parameters including adverse events | Baseline to Week 32
Incidence of safety parameters including abnormal laboratory results | Baseline to Week 32

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No